CLINICAL TRIAL: NCT04764877
Title: Effect of Osteopathic Manipulation Therapy on Pulmonary Function Testing in Children With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Alex Rakowsky, Assistant Professor Primary Care Pediatrics/Associate Residency Program Director, Nationwide Children's Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB #14-000667
Record Dates: First submitted 2021-01-21; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Asthma in Children
Keywords: OMM

STUDY DESIGN:
Intervention Model Description: Patients were randomized to either standard of care/teaching at our Hilltop Primary Care Center Asthma clinic OR to standard of care/teaching PLUS one time osteopathic manipulation focusing on improving lung expansion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Standard teaching and physical exam for any patient that would be seen at our Hilltop Primary Care center asthma clinic. This included baseline PFTs. FOR THIS STUDY a second set of PFTs were obtained at the end of the visit
- OMT arm (Experimental): As above BUT with the addition of standardized OMT focusing on lung functionality. OMT provided by either our OMM attending at that time (Dr Wolf) or residents trained by her for this study (Drs. Regan, Jones, Pe and Bryant)
  Interventions: Other: Osteopathic Manipulative Medicine

INTERVENTIONS:
Other: Osteopathic Manipulative Medicine — Provided 15-20 minute long OMT session for patients in the OMT arm
  Arms: OMT arm

SUMMARY:
Objective To evaluate change in same-day pulmonary function testing in pediatric patients receiving OMT compared to those receiving usual care.

Methods For this study, we selected patients utilizing the following inclusion criteria: 1) ages 7-18 years, 2) a diagnosis of asthma, 3) patients receiving care at a primary care-based asthma clinic, and 4) those patients who had baseline spirometry. Selected patients were then randomized to either an OMT or a control group. We excluded patients who were experiencing an acute asthma exacerbation. Patients in the OMT group were treated with rib raising and suboccipital release, in addition to standard asthma care, while control group patients received standard care only. A second PFT was performed on both groups at the end of the visit. OMT was performed by multiple osteopathic pediatric residents who were specifically trained for the purposes of this study. Change in spirometry results (FVC, FEV1, FVC/FEV1, and FEF 25-75%) were then compared.

DETAILED DESCRIPTION:
Objective To evaluate change in same-day pulmonary function testing in pediatric patients receiving OMT compared to those receiving usual care.

Methods For this study, we selected patients utilizing the following inclusion criteria: 1) ages 7-18 years, 2) a diagnosis of asthma, 3) patients receiving care at a primary care-based asthma clinic, and 4) those patients who had baseline spirometry. Selected patients were then randomized to either an OMT or a control group. We excluded patients who were experiencing an acute asthma exacerbation. Patients in the OMT group were treated with rib raising and suboccipital release, in addition to standard asthma care, while control group patients received standard care only. A second PFT was performed on both groups at the end of the visit. OMT was performed by multiple osteopathic pediatric residents who were specifically trained for the purposes of this study. Change in spirometry results (FVC, FEV1, FVC/FEV1, and FEF 25-75%) were then compared.

NOTE: The OMTs were done either by our OMM attending at that time (Dr. Wolf) or by residents trained by her for this study (Drs. Jones, Pe, Bryant and Regan,)

ELIGIBILITY:
Inclusion Criteria:

* Age as noted above
* Diagnosis of asthma
* Scheduled for routine asthma care at our clinic
* at least one prior PFT done prior to this visit

Exclusion Criteria:

* Clinical indication for pre- and post-bronchodilator spirometry on day of visit
* albuterol use w/in 8 hours of the visit
* oral steroid use in previous 2 weeks
* diagnosis of asthma exacerbation w/in prior 4 weeks

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in FEV1 on pre-therapy and post-therapy PFTs | 2 hours
  FEV1 improvement
Change in FEF25-75 on pre-therapy and post-therapy PFTs | 2 hours
  FEV25-75 improvement
Change in FVC on pre-therapy and post-therapy PFTs | 2 hours
  FVC improvement
Change in FVC/FEV1 on pre-therapy and post-therapy PFTs | 2 hours
  Improvement in ratio

SECONDARY OUTCOMES:
Standardized survey to look for adverse effects from the OMT | 2 hours
  Standard form asking about common AEs seen with OMT

IPD SHARING:
Plan to Share IPD: Yes
Study is completed and pending publication in the Journal of Osteopathic Medicine (formerly JAOA) Once published we do plan to share data with those interested
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication
Access Criteria: From interested OMT researchers